CLINICAL TRIAL: NCT06379074
Title: Poor Sleep During Pregnancy as Risk Factor for Post-partum Stress and Mental Health: A Translational, Longitudinal and Clinical Study. Maternal Outcome After THERapy for Sleep (MOTHERS)
Brief Title: Poor Sleep During Pregnancy as Risk Factor for Post-partum Stress and Mental Health
Acronym: MOTHERS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome G. Marconi (Other)
Collaborators: University of Bologna (Other); University of the Italian Switzerland (Other)
Responsible Party: Principal Investigator, Chiara Baglioni, Professor, University of Rome G. Marconi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022PMFMSE; C53D23004250008 (Other Grant/Funding Number: Italian Ministry of University and Research (MUR))
Record Dates: First submitted 2024-04-02; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Postpartum Depression; Insomnia; Stress
Keywords: Insomnia; Pregnancy; Stress; Sleep health; Postpartum; Actigraphy; Cortisol; DNA methylation; CBT-I
MeSH Terms: conditions — Depression, Postpartum; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants will receive a personal e-mail address to access their reserved area of the study's website. Each e-mail address is created using the pre-defined pseudonymized code, which will be assigned to each participant after screening (participants with sleep difficulties will be randomly assigned a code for condition B1 or B2).
  This procedure is designed to increase privacy protection, allow for matching of responses throughout study's phases, and blind outcome assessors to participants allocation.
  The personal website areas include contents based on their group allocation:
  * A: online questionnaire and sleep diaries;
  * B1: online questionnaire and sleep diaries; placebo intervention's contents (videos and pdf);
  * B2: online questionnaire and sleep diaries; intervention's contents (videos and pdf); weekly optional private chat with a clinician (a psychotherapist expert in CBT-I and insomnia during pregnancy).
Who Masked: Outcomes Assessor
Masking Description: Each participant will be assigned an identification code (ID-code) randomly generated by a computer. The codes associated to participants in Group B will be randomly assigned to intervention (Group B2) or placebo (Group B1). E-mail addresses will be created for each participant using the ID-code to access the private area of the study website. The code will be associated with responses to online questionnaires, actigraphy recording, saliva samples and sleep diaries.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subgroup B2: CBT-I derived intervention (Experimental): CBT-I derived intervention: 6 weekly online sessions with psychoeducation on sleep adapted to pregnancy, introduction of CBT-I techniques, discussion of sleep diaries and of acquired skills.
  Interventions: Behavioral: Improving sleep health and resilience during pregnancy
- Subgroup B1: psychological placebo intervention (Placebo Comparator): Psychoeducation placebo control intervention: 6 weekly online sessions composed of educational videos (ca. 20 minutes) on aspects related to pregnancy and sleep.
  Interventions: Behavioral: Information on pregnancy-related issues
- Group A: control group (No Intervention): A control group of healthy pregnant women with no insomnia complaints (ISI < 8) will be followed parallel to the intervention and control group, from the first trimester of pregnancy to 6 months post-partum to assess changes in sleep and psychological indices in pregnancy.

INTERVENTIONS:
Behavioral: Improving sleep health and resilience during pregnancy — Weekly sessions include: a video clip (ca. 20 min) and a pdf; short questions on participants' experience related to the session's content; brief feedback questions on session's contents. Participants will have weekly opportunity for private online chats with a clinician.
  Sessions' contents:
  1. Aims of the intervention; introducing the physiological regulation of sleep, sleep health and how sleep changes during pregnancy;
  2. Psychological regulation of sleep and the impact of behaviors on sleep regulation; introducing the basics of CBT-I behavioral techniques;
  3. Cognitive factors maintaining sleep difficulties; introducing cognitive techniques;
  4. Emotional factors maintaining sleep difficulties and on the bidirectional association between sleep and emotions; introducing emotion regulation techniques;
  5. Sleep in the postpartum and the development of sleep regulation in children;
  6. Relapse prevention and focus on acquired skills and how to prioritize sleep.
  Other Names: Sleeping for…2. Taking care of sleep during pregnancy and the post-partum
  Arms: Subgroup B2: CBT-I derived intervention
Behavioral: Information on pregnancy-related issues — Each session will include: video clip (ca. 20 minutes) on aspects related to pregnancy and sleep; brief feedback questions. Participants in the placebo intervention will not be given specific indications on skills or techniques for sleep difficulties and will not have access to the weekly chat with the clinician.
  Sessions will cover the following contents:
  Session 1: phases of pregnancy; Session 2: sleep disorders; Session 3: nutrition and physical activity during pregnancy; Session 4: childbirth; Session 5: psychophysical development of the child in the first three years of life; Session 6: synthesis of previous sessions.
  Other Names: Getting to know pregnancy ... pregnancy and postpartum information meetings
  Arms: Subgroup B1: psychological placebo intervention

SUMMARY:
Improving maternal mental health is a worldwide health priority. Nevertheless, several scientific sources highlighted lack of empirical data which could drive clinical practice. The present project addresses psychobiological mechanisms leading to peripartum mental disorders. It focuses on one key risk factor for psychopathology, which is poor sleep continuity. The project aims to describe the link between maternal poor sleep quality and the cascade of events which may enhance vulnerability to stress and risk for mental disorders and to evaluate the efficacy of an online automated psychological prenatal intervention directed to sleep problems in preventing these negative outcomes.

DETAILED DESCRIPTION:
The present trial aims to evaluate long-term effectiveness of a digital psychoeducational module based on CBT-I for expectant mothers complaining insomnia symptoms without psychiatric comorbidities on:

1. physiological, biological, genetical and subjective indices of maternal psychopathology, stress, and emotional processes. These outcomes will be assessed through online questionnaires and sleep diaries, cortisol levels, and recording of the sleep-wake activity through actigraphy;
2. father's and child's sleep and perceived stress. These outcomes will be assessed through online questionnaires and sleep diaries.

   114 expectant mothers will be evaluated from early pregnancy until 6 months post-partum.

   For power calculation of human studies, efficacy of clinical intervention for insomnia during pregnancy in preventing and ameliorating sleep, psychopathology and attachment with future child at post-partum was considered the primary outcome. A study that compared scores on the Edinburgh Postnatal Depression Scale (EPDS) in 132 women divided into cognitive-behavioral therapy for insomnia (N = 89) or control group (N = 43) before, during and after pregnancy was used. G-Power software estimated that 114 women in total would be needed to have an effect power of at least 80%.

   Women will be recruited primarily in the area of Bologna and Rome (Italy) and study's materials will be conserved in the Department of Biomedical and Neuromotor Sciences, University of Bologna (Italy).

   Screening: all interested women will be contacted for an appointment with a clinical psychologist for the screening, which will be conducted in a confidential space in a room at the Universities' Department involved (Department of Biomedical and Neuromotor Sciences, University of Bologna; Department of Human Sciences, Guglielmo Marconi University of Rome). These spaces will be used for all in-person contact with the participants (details below). Study's materials, including biological samples, will be conserved in a secured room in the Department of Biomedical and Neuromotor Sciences, University of Bologna for the whole duration of the study. All women will be asked to read and sign the informed consent before proceeding. Women will be evaluated through a widely used psychological structured interview (Structured Clinical Interview for DSM-5, SCID-5 in the brief version QuickSCID-5) and an interview about sleep. Furthermore, data on pregnancy and socioeconomic variables will be collected. Women will be asked to share, along with their consent, gynecological medical data on their health status (e.g. information on pregnancy). This face-to-face screening procedure will be conducted for checking inclusion criteria.

   The full sample will be divided in the following groups matched for age.
   1. Group A: control group of healthy pregnant women with no insomnia complaints (N=38);
   2. Group B: pregnant women complaining of subthreshold or clinical insomnia (N=76), further assigned to the following subgroups: Subgroup B1: psychological placebo intervention (N=38), Subgroup B2: CBT-I derived intervention (N=38).

   Insomnia complaints will be assessed through a validated questionnaire 'Insomnia Severity Index'. No insomnia complaints (Group A) vs insomnia complaints (Group B) will be operationalized using the cut-off of 7 (subthreshold insomnia). Group B will be randomly assigned to Subgroup B1 and to Subgroup B2.

   After the baseline interview, all women will be monitored longitudinally in 6 assessment evaluations:
   1. Baseline: between the 11th and the 15th week of pregnancy;
   2. Follow-up-1: after 6 weeks from baseline;
   3. Follow-up-2: after 12 weeks from baseline;
   4. Follow-up-3: 1-to-2-weeks after birth;
   5. Follow-up-4: 3-months post-partum;
   6. Follow-up-5: 6-monhts post-partum.

   For women who will be offered clinical treatment, baseline and follow-up-1 assessments will be conducted pre- and post-treatment.

   At three time points (Baseline, Follow-up 1, and Follow-up 5) an ecological-momentary-assessment (EMA) design will be used to collect data on sleep and emotions (sleep diary), sleep-wake parameters (actigraphy) and stress reactivity (salivary cortisol). Women will be asked, for each EMA week, to complete a sleep and emotion diary twice a day (in the morning and evening), to wear a wrist actigraph for 7 days, and to collect, on the first day of each EMA week, saliva samples through swabs. Saliva samples will be collected in the morning and the evening and will be used to evaluate salivary cortisol levels by liquid chromatography-tandem mass spectrometry (LC-MS/MS). Cortisol levels will be used as index of stress reactivity. Aliquots of morning salivary (1 assessment per person) will be used for the analysis of DNA methylation of the genes FKBP5, BDNF, and NR3C1, by Sequenom MALDI-TOF mass spectrometry, as potential biomarkers of prenatal poor sleep.

   The partner of each participant (n=114) will also be invited to take part to the study by filling out online questionnaire and sleep diaries for each assessment point detailed above.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 yrs. old;
2. good knowledge of Italian language;
3. intention to continue pregnancy;
4. BMI ranging 18-30 (i.e., without underweight or obesity following international criteria; WHO, 2013);
5. ≤ 15th week of pregnancy at the time of recruitment.

Exclusion Criteria:

1. severe diagnosis of relevant somatic disorder;
2. smoking;
3. alcohol intake;
4. assumption of illegal drugs;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2025-08-06 (Estimated); Study Completion 2025-10-06 (Estimated)

PRIMARY OUTCOMES:
Stress reactivity | Twice a day (morning and evening) once at baseline; after 6 weeks from baseline; 6 months post-partum
  Salivary cortisol level by saliva sample provided by participants through swab
Sleep efficiency | One week at baseline; after 6 weeks from baseline; 6 months post-partum
  Total Sleep Time (min)/Time In Bed (min) expressed in percentage and assessed through actigraphy monitoring
Depressive symptoms | Baseline; after 6 weeks from baseline; after 12 weeks from baseline; 1-to-2-week after birth; 3 months post-partum; 6 months post-partum
  Edinburgh Postnatal Depression Scale (EPDS) total score (min. = 0; max. = 30; higher scores indicate a greater probability of having depression)
Insomnia symptoms | Baseline; after 6 weeks from baseline; after 12 weeks from baseline; 1-to-2-week after birth; 3 months post-partum; 6 months post-partum
  Insomnia Severity Index total score (min. = 0; max. = 28; higher scores indicate a higher severity of insomnia)
Anxiety symptoms | Baseline; after 6 weeks from baseline; after 12 weeks from baseline; 1-to-2-week after birth; 3 months post-partum; 6 months post-partum
  Generalized Anxiety Disorder questionnaire total score (min. = 0; max. = 21; higher scores indicate a higher level of generalized anxiety)
Valence of affective states | Baseline; after 6 weeks from baseline; after 12 weeks from baseline; 1-to-2-week after birth; 3 months post-partum; 6 months post-partum
  Valence of morning and evening affective states assessed through visual scale in sleep and emotion diaries
Arousal of affective states | Baseline; after 6 weeks from baseline; after 12 weeks from baseline; 1-to-2-week after birth; 3 months post-partum; 6 months post-partum
  Arousal of morning and evening affective states assessed through visual scale in sleep and emotion diaries
Emotion regulation | Baseline; after 6 weeks from baseline; 6 monhts post-partum
  Cognitive Emotion Regulation Questionnaire - Italian Short-Version (each of the nine subscales' scores ranges from 2 to 10; higher scores indicate a greater use of a specific emotion regulation strategy)

SECONDARY OUTCOMES:
Mothers' parenting stress | 1-to-2-week after birth; 3 months post-partum; 6 months post-partum
  Parenting Stress Index-SF total and subscales score (subscales scores range from 12 to 60 and total score ranges from 36 to 180; higher scores indicate higher level of stress)
Partners' insomnia symptoms | Baseline; after 6 weeks from baseline; after 12 weeks from baseline; 1-to-2-week after birth; 3 months post-partum; 6 months post-partum
  Insomnia Severity Index total score (min. = 0; max. = 28; higher scores indicate a higher severity of insomnia)
Children sleep difficulties | 1-to-2-week after birth; 3 months post-partum; 6 months post-partum
  Brief Infant Sleep Questionnaire total score. Sleep difficulties are defined as: (1) the child wakings > 3 times per night; (2) the nocturnal wakefulness period > 1 h; or (3) the total sleep time < 9 h

OTHER OUTCOMES:
Partners' sleep efficiency | One week at baseline; after 6 weeks from baseline; 6 monhts post-partum
  Total Sleep Time (min)/Time In Bed (min) expressed in percentage and assessed through sleep diaries
Fathers' parenting stress | 1-to-2-week after birth; 3 months post-partum; 6 months post-partum
  Parenting Stress Index-SF total and subscales score (subscales scores range from 12 to 60 and total score ranges from 36 to 180; higher scores indicate higher level of stress)
Daytime sleepiness | Baseline; after 6 weeks from baseline; after 12 weeks from baseline; 1-to-2-week after birth; 3 months post-partum; 6 months post-partum
  Epworth Sleepiness Scale total score (min. = 0; max. = 24; higher scores indicate higher levels of sleepiness)

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Baglioni, Professor, Study Director — Department of Human Sciences, Guglielmo Marconi University, Rome, Italy
Locations (1):
- Department of Biomedical and Neuromotor Sciences, Physiology campus, University of Bologna, Bologna, Italy, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Austin MP, Frilingos M, Lumley J, Hadzi-Pavlovic D, Roncolato W, Acland S, Saint K, Segal N, Parker G. Brief antenatal cognitive behaviour therapy group intervention for the prevention of postnatal depression and anxiety: a randomised controlled trial. J Affect Disord. 2008 Jan;105(1-3):35-44. doi: 10.1016/j.jad.2007.04.001. Epub 2007 May 8. PMID 17490753
- [Background] First & Williams. QuickSCID-5. Raffaello Cortina Editore - Libro Raffaello Cortina Editore; 2020. https://www.raffaellocortina.it/scheda-libro/michael-b-first-janet-bw-williams/quickscid-5-9788832853629-3590.html
- [Background] Meneo D, Bacaro V, Buonanno C, Baglioni C. La valutazione del sonno in psicoterapia: una proposta di intervista clinica semistrutturata | Giovanni Fioriti Editore. Cognitivismo clinico. Published online November 9, 2023. https://www.fioritieditore.com/la-valutazione-del-sonno-in-psicoterapia-una-proposta-di-intervista-clinica-semistrutturata/
- [Derived] Meneo D, Baldi E, Cerolini S, Curati S, Bastianini S, Berteotti C, Simonazzi G, Manconi M, Zoccoli G, De Bartolo P, Gelfo F, Martire VL, Baglioni C. Promoting sleep health during pregnancy for enhancing women's health: a longitudinal randomized controlled trial combining biological, physiological and psychological measures, Maternal Outcome after THERapy for Sleep (MOTHERS). BMC Psychol. 2024 Jun 10;12(1):340. doi: 10.1186/s40359-024-01827-1. PMID 38858743